CLINICAL TRIAL: NCT02352233
Title: Pentax Retroview Colonoscope for the Evaluation of Colon Mucosa in Forward and Retro Viewing: a Safety and Feasibility Pilot Study
Brief Title: Retroview Colonoscope for the Evaluation of Colon Mucosa Study
Acronym: REVCOR
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: IECED 01-14-2014; IECED 2014-01 (Other: IECED 2014-01)
Record Dates: First submitted 2014-08-05; First posted 2015-02-02 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2014-09

CONDITIONS: Colonic Diseases
Keywords: retroview colonoscope; retroflexion colonoscopy; colonoscopy
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — biopsies, tissue from colonic mucosa: inflammatory, polyps
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- colonoscopy group: consecutive patients undergoing for colonoscopy for any formal indication. Patients were submitted to colonoscopy using RETROVIEW colonoscope
  Interventions: Procedure: RETROVIEW colonoscope

INTERVENTIONS:
Procedure: RETROVIEW colonoscope — withdrawal in retro vision and forward vision was performed by segments (right, transverse, left, sigmoid colon and rectum). Retroflexed therapeutics procedures were executed when needed.
  Other Names: Retro view colonoscopy; Retroflexion during colonoscopy

SUMMARY:
Colonoscopy is the "gold standard" technique for diagnosis and treatment of colonic lesions. Moreover, high definition colonoscopes (HD) associated to digital chromoendoscopy had shown better results regarding adenoma and polyps detection when compared to standard non HD scopes. However, evidence shows that during standard colonoscopy many lesions could be missed, including polyps, cancer and other kind of lesions. This could be correlated to many factors and recently reports show evidence that lesions behind the folds could be missed because the limitation of a forward view examination. Until know, a new auxiliary imaging device called "Third Eye Retroscope" had demonstrated more lesions detection during colonoscopy using a retro view, but with some limitations as absence of HD vision, the need of additional equipment and the fact the device occupies the accessory channel, limiting therapeutic efficiency. Recently a new HD colonoscope called "RETROVIEW" (PENTAX Medical) has been developed. It permits visualization of colonic mucosa in forward view, in retroflex view and allows for performance of diagnostic and therapeutics in a single colonoscope.

DETAILED DESCRIPTION:
Primary outcome:

To determine the safety and feasibility of the retro view during colonoscopy using RETROVIEW colonoscope. Safety was measured by the number of bleeding or perforation rates as adverse event during the procedure. Feasibility was measured by the number of cases that is possible to achieve a retroflexion in the colon Secondary outcome: withdrawal phase time and total procedure time.

ELIGIBILITY:
Inclusion Criteria:

* undergoing colonoscopy for colorectal neoplasia screening, for polyp surveillance, or for diagnostic workup including anemia, abdominal pain, constipation, abnormal imaging; and if they were able to understand and provide written consent for the procedure.

Exclusion Criteria:

* age <18; pregnancy, included history of colon resection, known inflammatory bowel disease, polyposis syndrome, radiation therapy to abdomen or pelvis, suspicion of chronic stricture potentially precluding complete colonoscopy, presence of diverticulitis or toxic megacolon, hemophilia and concurrent enrollment in another clinical investigation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients undergoing for colonoscopy at the Instituto Ecuatoriano de Enfermedades Digestivas
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety | 3 months
  The safety was measured by the number of cases with bleeding or perforation
Feasibility | 3 months
  The feasibility was measured determining the number of cases that was possible to perform a retro view by segments in the colon.

SECONDARY OUTCOMES:
Withdrawal colonoscopy phase | 3 months
  withdrawal colonoscopy phase time measured in minutes (excluding time taking in minutes in case of therapeutics)
Total procedure time | 3 months
  Total procedure time including retro view and forward view in minutes (excluding time taking in minutes in case of therapeutics)

OTHER OUTCOMES:
Number of lesions | 3 months
  number of lesions detected during the entire colonoscopy
Endoscopic Treatment | 3 months
  number of endoscopic therapeutic procedures in retro vision during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD, Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas, Guayaquil, Guayas, Ecuador

REFERENCES:
- [Background] Waye JD, Heigh RI, Fleischer DE, Leighton JA, Gurudu S, Aldrich LB, Li J, Ramrakhiani S, Edmundowicz SA, Early DS, Jonnalagadda S, Bresalier RS, Kessler WR, Rex DK. A retrograde-viewing device improves detection of adenomas in the colon: a prospective efficacy evaluation (with videos). Gastrointest Endosc. 2010 Mar;71(3):551-6. doi: 10.1016/j.gie.2009.09.043. Epub 2009 Dec 16. PMID 20018280